CLINICAL TRIAL: NCT03574714
Title: The Role of Extracellular pH on Spermatozoa's Directional Movement in Vitro
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 180614NU
Record Dates: First submitted 2018-06-20; First posted 2018-07-02 (Actual); Last update posted 2019-08-02 (Actual); Status verified 2018-06

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Extracellular pH — Extracellular pH gradient

SUMMARY:
The purpose of this research project is to determine whether or not the directional movement of spermatozoa is influenced by a pH gradient by examining spermatozoa in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Normal semen sample

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Males who come in to have their semen quality assessed.
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-09-28 (Actual)

PRIMARY OUTCOMES:
Directional Movement | 5 minutes
  Observing whether cells move towards alkaline or acidic

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No
The samples will be anonymous